CLINICAL TRIAL: NCT04662086
Title: COVID-19 Outpatient Pragmatic Platform Study (COPPS): A Pragmatic Multi-arm, Adaptive, Phase 2, Blinded, Randomized Placebo-controlled Platform Trial to Assess the Efficacy of Different Investigational Therapeutics in Reducing Time to Disease Resolution or Viral Load Cessation, as Compared to Standard Supportive Care in Outpatients With COVID-19
Brief Title: COVID-19 Outpatient Pragmatic Platform Study (COPPS) - Master Protocol
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COPPS-Master Protocol
Record Dates: First submitted 2020-12-08; First posted 2020-12-10 (Actual); Results first posted 2023-05-30 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Covid19
Keywords: Master Protocol; Outpatient
MeSH Terms: conditions — COVID-19 | interventions — acebilustat; camostat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acebilustat (Experimental): Participants are randomized to receive either active acebilustat or matching placebo for 28 days.
  Interventions: Drug: Acebilustat
- Camostat (Experimental): Participants are randomized to receive either active camostat or matching placebo for 10 days.
  Interventions: Drug: Camostat

INTERVENTIONS:
Drug: Acebilustat — 100 mg capsule administered orally once daily
  Arms: Acebilustat
Drug: Camostat — 200 mg (2 x 100 mg tablet) administered orally four times daily (800 mg total daily dose).
  Arms: Camostat

SUMMARY:
The overall objective of this study is to efficiently evaluate the clinical efficacy and safety of different investigational therapeutics among adults who have COVID-19 but are not yet sick enough to require hospitalization. The overall hypothesis is that through an adaptive trial design, potential effective therapies (single and combination) may be identified for this group of patients.

COVID-19 Outpatient Pragmatic Platform Study (COPPS) is a pragmatic platform protocol designed to evaluate COVID-19 treatments by assessing their ability to reduce viral shedding (Viral Domain) or improve clinical outcomes (Clinical Domain). To be included into the platform, every investigational product will collect data for both Domain primary endpoints. Individual treatments to be evaluated in the platform will be described in separate sub-protocols.

DETAILED DESCRIPTION:
The platform study allows investigational products with objectives either: evaluating viral shedding (Virology Domain); and COVID-19 related Clinical Outcomes (Clinical Domain).

The primary objective for investigational products within the Viral Domain is:

A. To evaluate the efficacy of each therapeutic intervention in addition to standard supportive care (SSC) compared with SSC in reducing viral shedding of SARS-CoV-2 virus in outpatients with COVID-19 disease.

The primary objective for investigational products within for the Clinical Domain is:

B. To evaluate the efficacy of each therapeutic intervention in addition to SSC as compared to SSC in improving sustained clinical outcomes in outpatients with COVID-19 disease.

Secondary objectives are:

1. The objective of the non-assigned domain an investigational product is under.

   1. If under Clinical Domain, reduction in viral shedding.
   2. If under Viral Domain, time to sustained resolution of symptoms.
2. To evaluate the efficacy of each therapeutic intervention in reducing SARS-CoV-2 related hospitalizations, ED visits, or death in outpatients with COVID-19 disease.
3. To assess the development of antibodies against SARS-CoV-2
4. To evaluate the safety and tolerability of each therapeutic intervention compared with placebo (supportive care).

ELIGIBILITY:
Inclusion Criteria:

1. Outpatient setting
2. Age ≥ 18 years and ≤ 80 years at the time of the assessment
3. Able and willing to understand the study, adhere to all study procedures, and provide written informed consent
4. Initial diagnosis of COVID-19 disease as defined by an FDA-cleared molecular diagnostic assay positive for SARS-CoV-2 with no more than 72 hours from the initial swab used in the diagnosis to the time of commencing informed consent.
5. At baseline, at least two symptoms should have mild or higher severity score, where at least one of the mild symptoms is not cough, fatigue, or loss of smell/taste OR at least one symptom has a moderate or higher severity score on the COVID Outpatient Symptom Scale (COSS).
6. Participant's COVID-19 related symptom onset occurred within 7 days prior to time of randomization.
7. Other inclusion criteria specific to the investigational product that may, in the eyes of the investigator, be deemed necessary.

Exclusion Criteria:

1. At screening, the participant needs to be admitted to the hospital or is being evaluated for potential admission.
2. Previous use of experimental drugs that may be active against COVID-19 in the eyes of the investigators.
3. Participant yields a positive urine pregnancy test at screening.
4. Participant is using adrenocorticosteroids (except topical or inhaled preparations or oral preparations equivalent to or less than 10 mg of oral prednisone) or immunosuppressive or immunomodulatory drugs (e.g., immunosuppressants, anticancer drugs, interleukins, interleukin antagonists or interleukin receptor blockers).

   NOTE: Treatment of study participants following institutional COVID-19 treatment policies or guidelines, including the use of immunomodulatory medications, is permitted. This excludes treatment with agents that have the potential for direct antiviral activity, including convalescent plasma and NO, and co-enrollment into other clinical studies that evaluate investigational agents for COVID-19.
5. Participant has a serious chronic disease (e.g., uncontrolled human immunodeficiency virus [HIV], cancer requiring chemotherapy within the preceding 6 months, and/or moderate or severe hepatic insufficiency).
6. Has renal insufficiency including severe renal impairment and ESRD and/or requiring hemodialysis or continuous ambulatory peritoneal dialysis (CAPD).
7. Has liver impairment greater than Child Pugh A.
8. Has a history of alcohol or drug abuse in the previous 6 months.
9. Has a psychiatric disease that is not well controlled where controlled is defined as: stable on a regimen for more than one year.
10. Has taken another investigational drug within the past 30 days.
11. Is deemed by the Investigator to be ineligible for any reason.
12. Additional exclusions may pertain to specific drugs as described in study-specific protocols.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2021-04-23 (Actual); Primary Completion 2022-05-03 (Actual); Study Completion 2023-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manisha Desai, PhD, Principal Investigator — Stanford University; Upinder Singh, MD, Principal Investigator — Stanford University; Yvonne Maldonado, MD, Principal Investigator — Stanford University; Chaitan Khosla, PhD, Principal Investigator — Stanford University; Haley Hedlin, PhD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - ValleyCare Medical Center, Pleasanton, California
  - Stanford University, Stanford, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bunning B, Hedlin H, Purington N, Sundaram V, Kapphahn K, Weng Y, Cunanan K, Maldonado Y, Singh U, Khosla C, O'Hara R, Nicolls M, Springman E, Parsonnet J, Rogers A, Levitt J, Desai M. The COVID-19 Outpatient Pragmatic Platform Study (COPPS): Study design of a multi-center pragmatic platform trial. Contemp Clin Trials. 2021 Sep;108:106509. doi: 10.1016/j.cct.2021.106509. Epub 2021 Jul 16. PMID 34274494
- [Result] Levitt JE, Hedlin H, Duong S, Lu D, Lee J, Bunning B, Elkarra N, Pinsky BA, Heffernan E, Springman E, Moss RB, Bonilla HF, Parsonnet J, Zamanian RT, Langguth JJ, Bollyky J, Khosla C, Nicolls MR, Desai M, Rogers AJ. Evaluation of Acebilustat, a Selective Inhibitor of Leukotriene B4 Biosynthesis, for Treatment of Outpatients With Mild-Moderate Coronavirus Disease 2019: A Randomized, Double-Blind, Placebo-Controlled Phase 2 Trial. Clin Infect Dis. 2023 Jul 26;77(2):186-193. doi: 10.1093/cid/ciad187. PMID 36996150
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants receive placebo for 10 or 28 days.
- Acebilustat: Participants receive acebilustat (100 mg/day) for 28 days.
- Camostat: Participants receive camostat (800 mg/day) for 10 days.
Period: Overall Study
Arm/Group | Placebo | Acebilustat | Camostat
Started | 60 | 60 | 2
Received Allocated Treatment | 59 | 59 | 2
Completed | 55 | 56 | 1
Not Completed | 5 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Acebilustat | Camostat | Total
Number analyzed (Participants) | 60 | 60 | 2 | 122
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (14) | 41 (13) | 29 (6) | 41 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 38 | 1 | 79
  Male | 20 | 22 | 1 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 14 | 1 | 29
  Not Hispanic or Latino | 45 | 46 | 1 | 92
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/Alaska Native | 0 | 1 | 0 | 1
  Asian | 5 | 5 | 0 | 10
  Native Hawaiian or other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 2 | 1 | 0 | 3
  White | 46 | 43 | 1 | 90
  More than one race | 1 | 2 | 0 | 3
  Unknown | 1 | 3 | 1 | 5
  Other | 3 | 5 | 0 | 8
  Missing | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 60 | 60 | 2 | 122
Viral Shedding [Mean (Standard Deviation); unit: cycles] — Cycle threshold (Ct) denotes how many PCR cycles are required before the SARS-CoV-2 viral RNA reached a detectable level. Higher Ct values correspond to lower viral copy numbers. For reference, Ct values of 20 correspond to ~2.12 x 106 viral copies per milliliter, while a Ct value of 40 is undetectable and is considered the lower limit of detection of this RT-PCR test for SARS-CoV-2.
  cycles | 21.2 (5.8) | 20.5 (6.4) | 30.8 (13.1) | 21.0 (6.3)

OUTCOME MEASURES:

1. Primary Outcome: For Viral Domain: Change in Viral Shedding
Description: Change in shedding of SARS-CoV-2 virus through day 10 attained from self-collected nasal swab. Viral load (nucleic acid) was assessed by RT-PCR Ct over time, and is reported here as the average change in Ct values per day. Cycle threshold (Ct) denotes how many PCR cycles are required before the SARS-CoV-2 viral RNA reached a detectable level. Higher Ct values correspond to lower viral copy numbers. For reference, Ct values of 20 correspond to ~2.12 x 106 viral copies per milliliter, while a Ct value of 40 is undetectable and is considered the lower limit of detection of this RT-PCR test for SARS-CoV-2.
Time Frame: 10 days
Population: Intent-to-treat analysis set
Measure: Mean (95% Confidence Interval); unit: cycles
Arm/Group | Placebo | Acebilustat | Camostat
Number analyzed (Participants) | 60 | 60 | 2
cycles | 1.6 [1.5 to 1.7] | 1.7 [1.6 to 1.7] | 1.0 [0.4 to 1.6]
Statistical Analysis 1: Comparison: Placebo vs Acebilustat; A generalized linear mixed effects model with parameterization was utilized to capture the difference in change in viral shedding at day 10 between treatment arms. SARS-CoV2 viral RNA CT values were transformed using a standard Reference curve; Test type: Other; p = 0.20, Linear mixed-effects regression model — A p-value of <0.05 would be considered statistically significant

2. Primary Outcome: For Clinical Domain: Time-to-sustained-resolution
Description: Time from randomization to sustained symptom resolution assessed over a 28-day period. Resolution is defined as the first day where no symptoms are self-reported on all succeeding days through and including day 28, not including sense of taste or smell, and defining recovery for fatigue and cough as mild or none.
Time Frame: 28 days
Population: Intent-to-treat analysis set
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo | Acebilustat | Camostat
Number analyzed (Participants) | 60 | 60 | 2
days | 26 [17.5 to NA] — Not calculable due to insufficient number of events | NA [22 to NA] — Not calculable due to insufficient number of events | NA [NA to NA] — Not calculable due to insufficient number of events
Statistical Analysis 1: Comparison: Placebo vs Acebilustat; A two-sided log rank test at the 0.04999 level of significance for the final analysis required 78 events (i.e., sustained symptom resolution) to provide 80% power to detect a hazard ratio of 1.91. Based on previous outpatient COVID-19 trials at Stanford, assumed placebo and treatment arm median time to symptom resolution of 10 and 5 days, respectively, for a total sample size of 120 patients. Participants with missing data lasting through Day 28 were censored on Day 28; Test type: Other; p = 0.07, Cox proportional hazards model — A p-value of <0.05 would be considered statistically significant; Two-sided Cox proportional hazards model adjusted for age, sex, and receipt of baseline receipt of monoclonal antibodies; Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.34 to 1.04]

3. Secondary Outcome: Time to Viral Cessation
Description: Defined as the time in days from randomization to the first of two consecutive negative RT-PCR results of self-collected nasal swabs.
Time Frame: 28 days
Population: Intent-to-treat analysis set.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo | Acebilustat | Camostat
Number analyzed (Participants) | 60 | 60 | 2
days | NA [NA to NA] — Not calculable due to insufficient number of events | NA [NA to NA] — Not calculable due to insufficient number of events | NA [NA to NA] — Not calculable due to insufficient number of events

4. Secondary Outcome: Time to First Resolution
Description: Defined as the first study day where no symptoms are self-reported, not including sense of taste or smell, and defining recovery for fatigue and cough as mild or none.
Time Frame: 28 days
Population: Intent-to-treat analysis set
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo | Acebilustat | Camostat
Number analyzed (Participants) | 60 | 60 | 2
days | 11.5 [7.75 to 18.25] | 14 [7 to 18] | NA [NA to NA] — Not calculable due to insufficient number of events
Statistical Analysis 1: Comparison: Placebo vs Acebilustat; Test type: Other; p = 0.05, Linear mixed-effects regression model; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.38 to 1.01]

5. Secondary Outcome: Time to Full Resolution
Description: Defined as the study day where no symptoms are first self-reported.
Time Frame: 28 days
Population: Intent-to-treat analysis set
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo | Acebilustat | Camostat
Number analyzed (Participants) | 60 | 60 | 2
days | 13 [8.75 to 17.5] | 15 [11 to 18] | NA [NA to NA] — Not calculable due to insufficient number of events
Statistical Analysis 1: Comparison: Placebo vs Acebilustat; Test type: Other; Hazard Ratio (HR) = 0.59, 95% CI 2-sided [0.34 to 1.01]

6. Secondary Outcome: Number of Participants With SARS-CoV-2 Related Hospitalizations, Emergency Department (ED) Visits, or Death in Outpatients With COVID-19 Disease.
Time Frame: 28 days
Population: Intent-to-treat analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Acebilustat | Camostat
Number analyzed (Participants) | 60 | 60 | 2
Participants
  Hospitalization | 0 | 1 | 0
  ED visit | 2 | 0 | 0
  Death | 0 | 0 | 0
Statistical Analysis 1: Comparison: Placebo vs Acebilustat; Difference in incidence of ED visits; Test type: Other; p = 0.21, Fisher Exact — A p-value of <0.05 would be considered statistically significant

7. Secondary Outcome: Number of Participants That Developed Antibodies to SARS-CoV-2
Time Frame: 28 days
Population: Participants with available antibody data are included in the analysis. No antibody results data were collected in the Camostat arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Acebilustat | Camostat
Number analyzed (Participants) | 55 | 53 | 0
Participants | 55 | 53 |

ADVERSE EVENTS:
Time Frame: Up to 35 days
Description: Safety Analysis Set: per protocol, the safety analysis was performed using the as-treated population and includes all patients who received study treatment. As pre-specified in the study protocol, any clinical events related to the progression of COVID-19 (except death) would not be considered adverse events.
Arm/Group | Placebo | Acebilustat | Camostat
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/59 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/59 | 0/2
Other Adverse Events (participants affected / at risk) | 3/59 | 1/59 | 0/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=59) | Acebilustat (N=59) | Camostat (N=2)
Nausea (Gastrointestinal disorders) | 3 | 1 | 0

LIMITATIONS AND CAVEATS:
This camostat arm did not meet its planned enrollment and did not achieve statistical power as specified in the protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan: Master Protocol (2021-09-21): https://cdn.clinicaltrials.gov/large-docs/86/NCT04662086/Prot_SAP_000.pdf
  • Study Protocol and Statistical Analysis Plan: Acebilustat Sub-Protocol (2021-09-21): https://cdn.clinicaltrials.gov/large-docs/86/NCT04662086/Prot_SAP_001.pdf
  • Study Protocol and Statistical Analysis Plan: Camostat Sub-Protocol (2021-09-21): https://cdn.clinicaltrials.gov/large-docs/86/NCT04662086/Prot_SAP_002.pdf